CLINICAL TRIAL: NCT04922398
Title: Ovarian Injection of PRP (Platelet -Rich Plasma) Vs Normal Saline in Premature Ovarian Insufficiency: A Randomized Controlled Trial
Brief Title: Ovarian Injection of PRP (Platelet -Rich Plasma) Vs Normal Saline in Premature Ovarian Insufficiency
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ahmed Saad (Other)
Collaborators: Hawaa Fertility Center (Other)
Responsible Party: Sponsor-Investigator, Ahmed Saad, Assistant professor of obstetrics & gynecology, Benha University
Organization: Benha University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Hawaa-9
Record Dates: First submitted 2021-05-19; First posted 2021-06-10 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Premature Ovarian Failure
Keywords: premature ovarian failure; poor responders; poor ovarian reserve; PRP
MeSH Terms: conditions — Primary Ovarian Insufficiency | interventions — Saline Solution; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: 60 patients with premature ovarian failure will be divided into 2 groups. The group A consists of 30 patients, who will receive a PRP (autologous platelet-rich plasma injection) with activation with calcium chloride. The group B consists of 30 patients, who will receive a normal saline inj. 0.9% Nacl.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: PRP group (Active Comparator): Preparation of PRP sample fro the patient own blood then the volume immediately above the erythrocyte layer was collected. Calcium gluconate in conc. 1:9 will be used as an activator. After activation, in a period less than 2 min, approximately 4 ml of the PRP will be injected into each ovary by TVUS.
  Interventions: Biological: platelet rich plasma
- Group B: saline group (Placebo Comparator): consists of 30 patients, who will receive 4 ml of a normal saline inj. 0.9% Nacl. then injected into each ovary by TVUS.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Biological: platelet rich plasma — blood will be withdrawn from the patient then separation of the platelet rich layer and then injection in the ovary
  Arms: Group A: PRP group
Drug: Normal saline — 0.9% normal saline will be injected in each ovary
  Other Names: saline
  Arms: Group B: saline group

SUMMARY:
60 cases with premature ovarian insufficiency will be randomized to either receive PRP or saline injection in their ovaries. Then follow up by hormonal & ultrasound & clinically to monitor any changes

DETAILED DESCRIPTION:
In this pilot study, 60 patients will be included. All patients will have a premature ovarian insufficiency (PORs) who meet at least two of the following three Bologna criteria.

The following data will be registered for all the cases: age, weight, height, menstrual history, previous pregnancies and their outcome, no. of living children and age of the youngest, history symptoms, married for how long, infertility duration and whether primary or secondary. Estimation of Antral Follicle Count (AFC) will be done for all the patients by transvaginal ultrasound (TVUS). Finally, a blood sample will be withdrawn for the following lab. Investigations: FSH, LH, E2, AMH, TSH, Prolactin before inclusion of the patients in the study.

A written consent form will be signed by all patients after complete explanation of the procedures and the expectations of the trial. Patients will be randomized into 2 groups (A& B). All will undergo a transvaginal intervention through an ovum pickup needle 17 G for the procedure. The group A consists of 30 patients, who will receive a PRP (autologous platelet-rich plasma injection) with activation with calcium chloride. The group B consists of 30 patients, who will receive a normal saline inj. 0.9% Nacl.

Sample preparation of the PRP:

According to the classification proposed by Ehrenfest, 4 different types of PRP are defined, depending on the content of cells and the presence of fibrin. In regards to the Classification of PRP in this case study, it is used as a commercial type of PRP with the lower concentration (2.5 x 3 times) system, Ycellbio PRP. The process will be carried out under strict aseptic conditions as well as optimum temperature regulations, i.e., 21-24°C. PRP will be prepared according to the manufacturer's guidelines. Draw 1 CC anticoagulant (sodium citrate) into a 20 CC syringe. Coat the inside walls of the syringe with the drawn anticoagulant. Then draw 14 CC blood under complete aseptic condition into a 20 CC syringe. Swing the syringe slowly to mix blood and anticoagulant well. Inject the blood slowly into the Ycellbio tube. Straighten the tube when the blood reaches the Y-funnel. Inject the blood into the Ycellbiotube to the appropriate level as indicated by the lines. Close the Ycellbio tube with silicon stopper using a forceps. Centrifuge at 3500 RPM at time 5 min. After the 5 min. spin, the Buffy coat is well visible. Twist the controller to adjust the height of buffy coat to the marked line. Twist the controller to adjust the height of buffy coat to the marked line. Prepare a 18 G ½ needle and a 3 CC syringe for PRP harvest. Open the silicone stopper using an alcohol soaked cotton. Extract 2.0 CC PRP while slowly swirling the needle in the area of the PRP into a 3 CC syringe. The same process is done for another 3 blood samples to have a total of 8 ml PRP to be used for both ovaries.

In the last step, the volume immediately above the erythrocyte layer will be collected. Calcium gluconate in conc. 1:9 will be used as an activator. After activation, in a period less than 2 min, approximately 4 ml of the PRP will be injected into each ovary by TVUS.

Monitoring & follow up:

The changes in the hormones at day 3 of the menstrual cycle: FSH, LH, estradiol, AMH will be closely monitored,after the application of the procedure in each group after 3 months. The investigators will also monitor the number of antral follicles & changes in the menstrual cycles & spontaneous ovulation before and after 3 months.

ELIGIBILITY:
Inclusion Criteria:

* PORs who meet at least two of the following three Bologna criteria
* AMH: 0.1-1 ng/ml.

Exclusion Criteria:

* ovarian insufficiency due to gonadal dysgenesis and -
* chromosomal abnormalities,
* immunoglobulin A deficiency,
* the use of anticoagulants,
* psychotropic medicaments,
* psychiatric disorders,
* carcinomas or
* a history of chronic pelvic pain.
* Women with present infection,
* haemoglobin lower than 11 g/L or
* platelets lower than 150 x 10ʒ/μL were excluded from the study.

Ages: 20 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — only in female patients
Enrollment: 60 (Estimated)
Dates: Start 2021-06-20 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
FSH hormonal changes | 3rd day of the 3rd menstrual cycle after the procedure
  The changes in the hormones at day 3 of the menstrual cycle: FSH monitored
vaginal ultrasound monitoring of the ovaries | 3rd day of the 3rd menstrual cycle after the procedure
  monitor the number of antral follicles.
clinical follow up | 3rd day of the 3rd menstrual cycle after the procedure
  changes in the menstrual cycle by history taking & questionnaire
LH hormonal changes | 3rd day of the 3rd menstrual cycle after the procedure
  serum LH at day 3 of the menstrual cycle
E2 hormonal changes | 3rd day of the 3rd menstrual cycle after the procedure
  serum E2 at day 3 of the menstrual cycle
AMH hormonal changes | 3rd day of the 3rd menstrual cycle after the procedure
  serum AMH

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed F Elsherbiny, phd.MD, Study Director — Professor of OB & GYN
Locations (1):
- Benha University, Banhā, Qalyubia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
the protocol the excel sheet
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 6 months
Access Criteria: 6 months